CLINICAL TRIAL: NCT04374370
Title: Severe Acute Respiratory Syndrome Coronavirus 2 of the Genus Betacoronavirus (SARSCoV2) Convalescent Plasma (CP) Expanded Access Protocol (EAP)
Brief Title: SARSCoV2 (COVID-19) Convalescent Plasma (CP) Expanded Access Protocol (EAP)
Status: No longer available | Type: Expanded Access
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1596191
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: COVID; SARSCoV2 Convalescent Plasma

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: SARSCoV2 Convalescent Plasma — Provide expanded access to SARSCoV2 convalescent plasma (EAP) collected from matched donors as described to patients with severe or life-threatening illness owing to COVID-19.

SUMMARY:
Convalescent plasma has been administered to treat different infectious diseases previously with some success. There is currently no approved and proven treatment options available for the novel coronavirus disease (COVID-19 virus). Some early data has shown a potential benefit in treating hospitalized patients who have tested positive for COVID-19 with convalescent plasma infusions of fresh plasma donated by fully recovered COVID-19 patients. The antibodies present in the recovered patients' plasma may be of benefit in helping critically ill and infected patients recover from the COVID-19 virus.

DETAILED DESCRIPTION:
Convalescent plasma has been administered to treat different infectious diseases previously with some success. There is currently no approved and proven treatment options available for the novel COVID-19 virus. Some early data has shown a potential benefit in treating hospitalized patients who have tested positive for COVID-19 with convalescent plasma infusions of fresh plasma donated by fully recovered COVID-19 patients. The antibodies present in the recovered patients' plasma may be of benefit in helping critically ill and infected patients recover from the COVID-19 virus. The purpose of this trial is to provide expanded access to SARSCoV2 convalescent plasma (EAP) collected from matched donors as described to patients with severe or life-threatening illness owing to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 and up
* Willing and able to provide written informed consent, or with a legal representative who can provide informed consent, or enrolled under International Conference on Harmonization (ICH) E6(R2) 4.8.15 emergency use provisions as deemed necessary by the investigator (participants ≥ 18 years of age); or willing and able to provide assent as required per Institutional Review Board (IRB) prior to performing study procedures.
* Must have laboratory confirmed COVID-19 positive test
* Must have severe or immediately life-threatening COVID-19

Severe disease is defined as:

1. dyspnea
2. respiratory frequency ≥ 30/min
3. blood oxygen saturation ≤ 93%
4. partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or
5. lung infiltrates > 50% within 24 to 48 hours

   Life-threatening disease is defined as:
6. respiratory failure
7. septic shock, and/or
8. multiple organ dysfunction or failure

Exclusion Criteria:

* Known contraindication to transfusion or history of prior reactions to transfusion of blood products

Ages: 6 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Oliveira, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

REFERENCES:
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428